CLINICAL TRIAL: NCT00700921
Title: Lovastatin as a Potential Modulator of Apoptosis in COPD
Brief Title: Lovastatin as a Potential Modulator of Apoptosis in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NJMRC HS-2163; NIH grant #HL088138
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Drug (Lovastatin) (Experimental)
  Interventions: Drug: Lovastatin
- Placebo (inactive comparator) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovastatin — 40mg po once daily
  Arms: Active Drug (Lovastatin)
Drug: Placebo — One capsule, once daily
  Arms: Placebo (inactive comparator)

SUMMARY:
This study will test whether lovastatin helps to modify lung inflammation in patients with COPD (Chronic Obstructive Pulmonary Disease).

DETAILED DESCRIPTION:
The impact of lovastatin, 40mg by mouth once daily on biological and clinical outcomes will be evaluated in an exploratory 16-week comparative treatment efficacy trial in 44 adult former smokers with established COPD of moderate severity. This trial employs a longitudinal randomized, parallel-arm, double-blind, placebo-controlled design using biomarkers of airway inflammation as the primary outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥45 years) former smokers with ≥ 10 pack-years of cigarette smoking
2. FEV1/FVC ratio < 70%
3. Post-bronchodilator FEV1 between 50% and 80% of predicted if undergoing bronchoscopy, or between 30% and 80% of predicted if undergoing induced sputum only
4. DLco/VA < 80% predicted
5. Ability to perform and adhere to study protocol
6. ability to provide informed consent.

Exclusion Criteria:

1. Asthma or other comorbid lung disease,
2. Hypoxemia (PaO2 < 55 mmHg or SpO2 < 88% on room air), if undergoing bronchoscopy
3. Exacerbation of COPD within the last 6 weeks
4. Upper or lower respiratory tract infection within the last 6 weeks
5. Current smoking
6. Significant coronary artery disease as reflected by unstable angina, myocardial infarction or angioplasty/stenting/bypass surgery within 6 months
7. Current use of HMG-coA-reductase inhibitors
8. Current use of inhaled corticosteroid
9. Concurrent use of other Cyp3A4 (isoform of cytochrome P450) inhibitors
10. History of adverse reaction to HMG-coA-reductase inhibitors (rhabdomyolysis, hepatitis)
11. For patients undergoing bronchoscopy, any contraindication to fiberoptic bronchoscopy or conscious sedation, including abnormalities of the platelet count, prothrombin time or partial thromboplastin time.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To determine the effects of lovastatin on apoptosis and efferocytosis in pulmonary macrophages. | 5 years

SECONDARY OUTCOMES:
To determine the effects of lovastatin on COPD phenotypic variables including lung function, exercise performance, clinical status and quality of life. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: E Rand Sutherland, MD, MPH, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No